CLINICAL TRIAL: NCT03963752
Title: Evidence-based Medical Research on the Treatment of Children's Rapid Progressive Central Precocious Puberty With Integrative Chinese and Western Medicine
Brief Title: Clinical Trial of Rapid Progressive Central Precocious Puberty With Integrative Chinese and Western Medicine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jian Yu, Director of TCM Department, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18401902300
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Idiopathic Precocious Puberty
Keywords: Idiopathic Precocious Puberty; Rapid Progressive; Integrative Chinese and Western Medicine; Evidence-based Medicine
MeSH Terms: interventions — Megestrol Acetate; Leuprolide; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ziyinxiehuo Granules and Megestrol Acetate (Experimental): Experimental：Group Ziyinxiehuo Granules and Megestrol Acetate Tablet Intervention :Subjects in Group Ziyinxiehuo Granules and megestrol acetate tablet will be treated with Ziyinxiehuo Granules and megestrol acetate tablet for 6 months.1 pack of Ziyinxiehuo granules Herbs includes shengdi 5g, xuanshen 3g, zexie 3g, zhimu3g, huangpai 3g, zhiguiban 2g, maiya 6g,tiandong 3g, zhigancao 2g. Ziyinxiehuo Granules is administered after dissolved,1pack every time, 2 times per day after a meal; and the dosage of megestrol acetate is 6-8mg/d, which is taken in 3 times after a meal.
  Interventions: Drug: Ziyinxiehuo Granules Herbs; Drug: Megestrol Acetate Tablet
- Gonadotrophin (Active Comparator): Active Comparator: Group Gonadotrophin Intervention: Subjects in Group Gonadotrophin will be treated with gonadotrophin releasing hormone agonist for 6months. In our study Leuprorelin Acetate 3.75mg Injection will be applied, the dosage of which is 80μg/kg every time by subcutaneous injection, every 4 weeks for once.
  Interventions: Drug: Leuprorelin Acetate 3.75mg Injection

INTERVENTIONS:
Drug: Ziyinxiehuo Granules Herbs — 1 pack of Ziyinxiehuo granules Herbs is administered after dissolved, 2 times per day after a meal.
  Other Names: nourishing"Yin"-removing"Fire" Granules
  Arms: Ziyinxiehuo Granules and Megestrol Acetate
Drug: Megestrol Acetate Tablet — the dose is 6-8mg/d, three times per day after meals.
  Arms: Ziyinxiehuo Granules and Megestrol Acetate
Drug: Leuprorelin Acetate 3.75mg Injection — Usage： 80μg/kg by subcutaneous injection, every 4 weeks
  Arms: Gonadotrophin

SUMMARY:
Our study used a randomized controlled trial to validate the clinical efficacy of a combination of traditional Chinese and Western medicine in the treatment of children with rapid progressive central precocious puberty.

DETAILED DESCRIPTION:
In the research, 164 subjects diagnosed with rapid progressive idiopathic precocious puberty are randomly divided into Group Ziyinxiehuo Granules and Megestrol Acetate Tablet（82 cases）and Group Gonadotrophin ( 82 cases). Patients in Group Ziyinxiehuo Granules and Megestrol Acetate Tablet are treated with ziyinxiehuo Granules and megestrol acetate tablet , whereas the Group Gonadotrophin received with gonadotrophin releasing hormone agonist, and all the subjects in two groups are continuously treated for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Girls are diagnosed as Idiopathic central precocious puberty by GnRH （gonadotrophin releasing hormone）Stimulation Test, and their age of onset ≤8 years;
* Tanner stages of breast in female patients ≥ Tanner III stage，diameter of mammillary nucleus ≥ 3cm;
* B-type ultrasonography: the volume of uterus≥3ml, the volume of ovary≥1.5ml, the diameter of follicle≥4mm;
* Bone age: compared the chronological age, the bone age is more than 1 year and the bone age <11.5 years old;
* It progresses rapidly, ratio of bone age difference to chronological age difference> 1;
* No GnRH analogs or sex hormones were administrated in the past;
* All above are needed at the same time.

Exclusion Criteria:

* Precocious precocity caused by the central nervous system organic diseases;
* Precocious precocity caused by congenital hypothyroidism, congenital adrenal hyperplasia, adrenal tumor and ovarian or testicular neoplasms as well as McCune-Albright syndrome, etc;
* Precocious precocity with a family history of diseases such as tumor, leukemia, diabetes, systemic lupus erythematous;
* Pseudo sexual precocity and partial precocious puberty.

Ages: 5 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of the Mammary Nucleus Diameter reduced to less than 1cm | After six months of continuous treatment
  The investigators will measure subjects' mammary nucleus diameter through the midline of the breast with a ruler after six months of continuous treatment, and percentage of the mammary nucleus diameter reduced to less than 1cm in each group will be calculated.

SECONDARY OUTCOMES:
Ratio of bone age difference to chronological age difference | After six months of continuous treatment
  The left hand orthotopic X-ray (including the carpal bone and the lower end of the ulna) will be filmed by the Department of Radiology before and after treatment, and the bone age will be measured according to the Greulich-Pyle map method. Ratio of bone age difference to chronological age difference will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yu, professor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No